CLINICAL TRIAL: NCT07025655
Title: The Effectiveness of a Multifaceted Mindfulness Program Integrated With Digital Technology-Assisted Learning on Healthy Aging in Community-Dwelling Older Adults: A Randomized Controlled Trial
Brief Title: Effectiveness of a Mindfulness and Digital Technology Program for Healthy Aging (MMP-DTLA)
Acronym: MMP-DTLA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University of Science and Technology (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Yu-Rung Wang, Assistant Professor, Chang Gung University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202400087B0C6001; NSTC 113-2410-H-255 -001 -MY2 (Other Grant/Funding Number: National Science and Technology Council of Taiwan)
Record Dates: First submitted 2025-04-30; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-04

CONDITIONS: Mindfulness; Healthy Aging
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental): Ten-week mindfulness programs supported by digital technology-assisted teaching materials
  Interventions: Behavioral: Multifaceted Mindfulness Program
- Control (Placebo Comparator): No intervention
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Multifaceted Mindfulness Program — Ten-week mindfulness classes
  Other Names: Mindfulness
  Arms: Mindfulness
Behavioral: Placebo — Regular daily activity
  Arms: Control

SUMMARY:
This study aims to evaluate the effectiveness of a mindfulness program integrated with digital technology-assisted learning on healthy aging among community-dwelling older adults. In a randomized controlled trial, 100 participants will be randomly assigned to either an experimental or a control group. The experimental group will receive a ten-week mindfulness program supported by digital tools such as educational videos and LINE Bot messaging. Primary outcomes include mindfulness awareness, physical activity, heart rate variability, cognitive function, sleep quality, perception of aging, and healthy aging perspectives. Additionally, qualitative interviews will be conducted with 10 experimental group participants to explore their intervention experiences.

ELIGIBILITY:
Inclusion Criteria:

1. ability to communicate in Mandarin or Taiwanese
2. aged 65 years or older in the community
3. Currently using a mobile phone and the LINE application as a means of communication.

Exclusion Criteria:

* Individuals with cognitive impairments
* Unable to communicate verbally

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-11 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
mindfulness awareness | We will collect four times of data: 1. Baseline 2. The fourth week 3. Up to 10 weeks 4. After completing the study for one month
  The Five Facet Mindfulness Questionnaire (FFMQ) will be used. Items are rated on a 5-point Likert scale ranging from 5 (almost always) to 1 (never), with higher scores indicating greater frequency. Certain items are reverse-coded, and total scores are computed after adjusting for these items. A higher total score reflects a greater level of mindfulness.
Physical activity: PASE-C | We will collect four times of data: 1. Baseline 2. The fourth week 3. Up to 10 weeks 4. After completing the study for one month
  The PASE-C encompasses domains including total physical activity, leisure activities, household activities, and occupational activities. Higher scores indicate greater levels of physical activity.
Physical activity: SPPB | We will collect four times of data: 1. Baseline 2. The fourth week 3. Up to 10 weeks 4. After completing the study for one month
  The SPPB comprises three components: balance tests, gait speed tests, and chair stand tests. A total score ranging from 0 to 9 indicates mobility impairment, whereas a score between 10 and 12 reflects normal mobility function.
Cognitive function | We will collect four times of data: 1. Baseline 2. The fourth week 3. Up to 10 weeks 4. After completing the study for one month
  The Montreal Cognitive Assessment (MoCA) will be used to assess cognitive function among community-dwelling older adults. The total score ranges from 0 to 30, with higher scores indicating better overall cognitive functioning. A score of 26 or above is generally considered within the normal range.
Heart rate variability: SDNN | We will collect four times of data: 1. Baseline 2. The fourth week 3. Up to 10 weeks 4. After completing the study for one month
  Heart rate variability (HRV) was assessed using a monitoring device to evaluate autonomic nervous system activity. The standard deviation of normal-to-normal intervals (SDNN) reflects the variability in RR intervals from electrocardiogram recordings, with higher SDNN values indicating greater heart rate variability.
Heart rate variability: LF/HF ratio | We will collect four times of data: 1. Baseline 2. The fourth week 3. Up to 10 weeks 4. After completing the study for one month
  Heart rate variability (HRV) was assessed using a monitoring device to evaluate autonomic nervous system activity. Sympathetic and parasympathetic activity were assessed through frequency-domain measures, including low-frequency (LF) and high-frequency (HF) components. The LF/HF ratio was calculated to evaluate the balance of autonomic nervous system activity.
Sleep quality | We will collect four times of data: 1. Baseline 2. The fourth week 3. Up to 10 weeks 4. After completing the study for one month
  The study utilized the Pittsburgh Sleep Quality Index (PSQI) to measure sleep quality. The Pittsburgh Sleep Quality Index (PSQI) yields a global score ranging from 0 to 21, with higher scores indicating poorer sleep quality. A global PSQI score greater than 5 is indicative of clinically significant sleep disturbance.
Perception of ageing | We will collect four times of data: 1. Baseline 2. The fourth week 3. Up to 10 weeks 4. After completing the study for one month
  The perception of ageing was measured using the Brief Aging Perceptions Questionnaire (B-APQ). A 5-point Likert scale was used for scoring, with 1 indicating 'strongly disagree,' 2 'disagree,' 3 'neutral,' 4 'agree,' and 5 'strongly agree.' Higher scores reflect more positive perceptions of aging.
Healthy ageing perspectives | We will collect four times of data: 1. Baseline 2. The fourth week 3. Up to 10 weeks 4. After completing the study for one month
  The Healthy Aging Perspectives Questionnaire (HAPQ) will be used. This questionnaire adopts a 5-point Likert scale, where 1 indicates 'strongly disagree,' 2 'disagree,' 3 'neutral,' 4 'agree,' and 5 'strongly agree.' Higher scores indicate more positive perspective of healthy aging.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Rung Wang, PhD, Principal Investigator — Chang Gung University of Science and Technology, Chiayi Campus

IPD SHARING:
Plan to Share IPD: Undecided
This is for the participants' privacy and research ethics.

REFERENCES:
- [Background] Wang YR, Lee HF, Hsieh PL, Chang CH, Chen CM. Relationship between physical activity and perceptions of ageing from the perspective of healthy ageing among older people with frailty with chronic disease: a cross-sectional study. BMC Nurs. 2023 Sep 16;22(1):319. doi: 10.1186/s12912-023-01481-9. PMID 37716946
- See also: Using the mindfullness practice for the development of the program — https://www.randomhousebooks.com/books/89149/